CLINICAL TRIAL: NCT05897671
Title: Foveal Sparing ILM Peeling With ILM Flap Transposition
Status: Completed | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of department, Vienna Institute for Research in Ocular Surgery
Other Study IDs: FSI
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Full Thickness Macular Hole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: retrospective data analysis of patients that underwent after foveal sparing ILM peeling with ILM flap transposition for macular hole repair
  Interventions: Other: retrospective data analysis

INTERVENTIONS:
Other: retrospective data analysis — Macular hole closure rate, visual acuity and OCT

SUMMARY:
Foveal sparing internal limiting membrane (ILM) peeling with ILM flap transposition over the macular hole combines the benefits of foveal sparing ILM peeling with ILM flap techniques.

Aim of this study is to retrospectively examine the rate of postsurgical macular hole closure, development of central atrophy in the foveal area, and improvement of best corrected distant visual acuity in a group of patients having undergone foveal sparing ILM peeling with ILM flap transposition for macular hole repair.

DETAILED DESCRIPTION:
Idiopathic full thickness macular holes lead to central defects in the visual field and to deterioration of the visual acuity. Introduction of internal limiting membrane (ILM) Peeling techniques lead to significant increase in closure rates of the macular holes.

Foveal sparing ILM peeling represents a surgical technique for macular hole repair with less surgical trauma with high closure rates of the macular hole, compared to classic ILM Peeling [Ho et al. 2014, Murphy et al 2019]. The combination of foveal sparing ILM Peeling with the established ILM flap techniques [Michalewska et al 2010 und 2015] offers the potential of better improvement in postsurgical visual acuity with the high closure rates, due to ILM flaps.

Aim of this study is to retrospectively examine the rate of postsurgical macular hole closure, development of central atrophy in the foveal area, and improvement of best corrected distant visual acuity in a group of patients having undergone foveal sparing ILM peeling with ILM flap transposition for macular hole repair.

ELIGIBILITY:
Inclusion Criteria:

* Vitrectomy with foveal sparing ILM peeling with ILM flap transposition in the time period from 1.10.2020 to 8.7.2022
* Age 18 and older
* Idiopathic full thickness macular hole as indication for surgery
* Full follow-up, including visual acuity testing and OCT preoperative, and 3 months after surgery.

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be selected by the clinical investigators in the Hanusch Hospital
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
macular hole closure rate | up to 3 months after surgery
  postsurgical closure of macular holes is examined from routine postsurgical optical coherence tomography (OCT) imaging

SECONDARY OUTCOMES:
visual acuity | 3 months
  visual acuity before and 3 months after surgery is examined
OCT | 3 months
  measurements of macular hole diameters from presurgical OCTs and restoration of the ellipsoid zone (EZ) 3 months after surgery is analysed

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Principal Investigator — head of departement
Locations (1):
- Hanusch Hospital, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No